CLINICAL TRIAL: NCT07265453
Title: A Family Centred Approach to Enhance Lifestyle Change and Behavioural Modification for Prevention of Cardiovascular Diseases Among Adolescents and Their Families in Uganda
Brief Title: A Family-centred Approach Enhancing Cardiovascular Health in Ugandan Adolescents and Their Families
Acronym: FaCe-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: University of California (Other); The AIDS Support Organization (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RGJB230801
Record Dates: First submitted 2025-08-09; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior; Lifestyle Modification; Cardiovascular Disease Other
Keywords: cardiovascular risk; CVD; Ideal cardiovascular health; physical activity diary; food diary; diet diary; family centered
MeSH Terms: conditions — Adolescent Behavior | interventions — Therapeutics; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FaCe-D Control arm (Active Comparator)
  Interventions: Other: Control Arm - standard of care
- FaCe-D Intervention (Experimental): Family-centred approach for lifestyle changes and behavioural modification
  Interventions: Behavioral: The immediate (treatment) arm, will receive the FaCe-D intervention comprising of 'HOME VISITS, DIET, PHYSICAL ACTIVITY AND HEALTH MESSAGING

INTERVENTIONS:
Behavioral: The immediate (treatment) arm, will receive the FaCe-D intervention comprising of 'HOME VISITS, DIET, PHYSICAL ACTIVITY AND HEALTH MESSAGING — The participants will receive the FaCe-D intervention comprising of dietary and exercise interventions delivered by Village Health Teams (VHTs)
  Arms: FaCe-D Intervention
Other: Control Arm - standard of care — Arm Description: They will continue to receive standard care with VHts performing their usual roles of health promotion for both communicable and non-communicable diseases as outlined by the Ministry of Health guidelines. This standard care involves visits by the VHT at least once a quarter to check hygiene and environment, children's immunisation status and other health promotion activities. The VHT may or may not involve the entire family/household.
  Arms: FaCe-D Control arm

SUMMARY:
The FaCe-D Study, with funding from the Canadian Institute for Health Research (CIHR) through Global Alliance for Chronic Diseases (GACD) aims to adapt and implement an evidence-based family centred approach (FCA) to prevent cardiovascular diseases (CVD) among adolescents and their families. This 5-year implementation science study will be conducted in 16 villages in Jinja district and another 16 in Kampala beginning April 2024 to evaluate the effectiveness of FCA in reducing the risk of CVD in Uganda and to assess feasibility, adoption, while measuring the costs of implementation. The study will be implemented by a group of researchers from MRC/UVRI & LSHTM, University of British Columbia (Canada), TASO (Uganda) and University of California San Francisco (UCSF) - USA with guidance from the Ministry of Health - Uganda.

DETAILED DESCRIPTION:
Uganda faces a growing challenge of non-communicable diseases (NCDs) alongside the existing burden due to HIV/AIDS. By NCDs, the investigators refer to common conditions such as diabetes, cancers, and cardiovascular diseases (including hypertension, stroke, and heart attack). About 38.8% of the population in Uganda has raised blood pressure (pre-hypertension), 34% in urban and 22% in rural areas have hypertension. The risk factors, such as unhealthy diet and physical inactivity, responsible for the development of these NCDs are modifiable and related to behaviour. The investigators propose to adapt, implement and evaluate a family-centred approach to enhance behaviour change among adolescents and their families.

Why focus on Adolescents? The investigators recognize that adolescence is a critical stage marked by significant physical, cognitive, and social changes and time to adopt behaviour that extends into adulthood. Previous studies have shown that even if the signs and symptoms of cardiovascular disease appear in adulthood, the process starts earlier during adolescence. The investigators aim to intervene by working with adolescents and families to change their behaviors and adopt a healthier diet and engage in recommended level of physical.

The iHealth T2D study that was conducted in parts of Asia and the United Kingdom showed that using the family centered approach and working closely with community health care workers led to reduction in body weight, blood pressure and thus reducing the risk of NCDs among the Asian population. The investigators will adapt the iHealth T2D study intervention to the Ugandan context, considering the specific features of the setting, village health team responsibilities and content of the education material. The intervention will promote physical activity and healthy eating habits among families.

The study comprises three phases; a) formative phase which is focusing on adapting the intervention, b) Implementation phase, to implement the adapted intervention and c) evaluation phase, assessing effectiveness and the overall process of the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 -19 years
* Household head/parent has provided consent/permission
* Planning to continue staying in the study village for the next 12 months

Exclusion Criteria:

* In a boarding school or planning to join a boarding school
* Pregnant or lactating
* Known to have a chronic condition such as mental illness
* The adolescent does not assent or consent

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1280 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Ideal cardiovascular health | after 12 months of follow-up
  Ideal cardiovascular health (ICH) will be determined by the total score on the American Heart Association's 'Life's Simple 7' tool. The score ranges from 0 to 7 points, where a higher score represents better cardiovascular health.

SECONDARY OUTCOMES:
sleep quality | 12 months
  Sleep quality will be measured using the Single-Item Sleep Quality Scale (SQS) by Snyder et al. (2018). Participants will report their sleep quality over a 7-day recall period using a 10-point visual analogue scale, where 0=terrible and 10=excellent. Higher scores on the scale indicate better sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Rachel King, PhD, Principal Investigator — University of California, San Francisco; Prof David Moore, PhD, Principal Investigator — University of British Columbia; Dr Josephine Birungi, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (2):
- Uganda (2):
  - TASO Jinja, Jinja
  - Kiswa Health center III, Kampala

IPD SHARING:
Plan to Share IPD: Yes
Before data is made available, it will be deidentified
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the publication of the main results with no end date
Access Criteria: A link shall be provided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT07265453/Prot_SAP_000.pdf